CLINICAL TRIAL: NCT05345587
Title: Quality of Life and Economic Repercussions of Combining Proactive Medication Assessment and Electronic Monitoring of Toxicities in Subjects Undergoing Oral Cancer Therapy
Acronym: PROLIFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHRC-I/2019/FF-01
Record Dates: First submitted 2022-03-11; First posted 2022-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prolife group (Experimental): scheduled consultation with the hospital clinical pharmacist, therapeutic follow-up and collection of clinical information by the patient via the THESS monitoring system
  Interventions: Other: THESS monitoring
- Standard care (No Intervention)

INTERVENTIONS:
Other: THESS monitoring — Consultation with the pharmacist to look for possible medication interactions between the oral therapy and the patient's usual treatments and to inform the patient about his treatment to improve QOL and compliance. Consultation and follow-up by a nurse. Weekly notification by THESS Application of the symptoms experienced by the patient over the last 7 days
  Arms: Prolife group

SUMMARY:
Therapies used to treat cancer are administered orally (OT) in 75% of cases, lending themselves to outpatient care. This care pathway raises new issues: specific toxicities, drug interactions, and the relationship between the community (physicians and pharmacists) and the hospital.

Drug interactions can increase toxicities or decrease the effectiveness of treatment and impact overall survival. Detection of drug interactions before treatment initiation is not always performed in routine practice. However, these oral treatments have a low therapeutic index and are associated with side effects that can alter quality of life (QoL). They are classically documented by the physician at the time of the consultation using the Common Terminology Criteria for Adverse Events (CTCAE), which makes it possible to adapt management. Nevertheless, numerous studies have shown a discrepancy between side effects reported by the patient versus those recorded by the physician, who tends to underestimate the intensity of the effects experienced by the patient.

Studies have shown an improvement in the overall survival and QoL of patients followed by electronic patient reported outcomes (ePRO) compared to patients followed conventionally.

Therefore, for this study, the study investigators aim to measure the impact of a care pathway associating a scheduled consultation with the hospital clinical pharmacist integrating a proactive medication assessment and the search for drug interactions and a follow-up of toxicities by ePROs on the QoL of patients treated with oral therapies in oncology and to estimate the economic impact.

ELIGIBILITY:
Inclusion Criteria:

* Patient starting oral therapy treatment in oncology for metastatic or locally advanced cancer
* Patient able to use a connected electronic object
* Patient with a smartphone/tablet or computer with internet access and an email address.
* Patient with WHO status ≤2
* Patients receiving other cancer therapy concurrently with oral therapy may be included
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in a category 1 interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Patient pregnant, parturient or breast feeding
* Illiterate patient
* Patients with poor prognosis due to a serious uncontrolled medical condition, mild systemic disease, uncontrolled infection (cardiac, pulmonary, renal, etc.)
* Patient receiving hormone therapy alone for breast or prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time until decrease in quality of life by 5-points between groups | End of follow-up maximum 18 months
  Quality of life calculated every 3 months using EORTC QLQ-C30 for which a decrease of 5-points is considered to be the minimal clinically important difference

SECONDARY OUTCOMES:
Time until progression of cancer between groups | End of follow-up maximum 18 months
  Measured every 3 months by the Response Evaluation Criteria in Solid Tumours (RECIST) criteria, classed as: Complete response (CR), Partial response (PR), Stable disease (SD), or Progressive disease (PD)
Patient satisfaction with their treatment between groups | 3 months
  The EORTC PATSAT-C33 questionnaire assesses the delivery of oncology care as a whole with a score from 1-5; the EORTC OUT-PATSAT7 is a complementary questionnaire to assess the delivery of ambulatory oncology care with a score from 1-5.
Patient satisfaction with their treatment between groups | 6 months
  The EORTC PATSAT-C33 questionnaire assesses the delivery of oncology care as a whole with a score from 1-5; the EORTC OUT-PATSAT7 is a complementary questionnaire to assess the delivery of ambulatory oncology care with a score from 1-5.
Patient satisfaction with their treatment between groups | 9 months
  The EORTC PATSAT-C33 questionnaire assesses the delivery of oncology care as a whole with a score from 1-5; the EORTC OUT-PATSAT7 is a complementary questionnaire to assess the delivery of ambulatory oncology care with a score from 1-5.
Patient satisfaction with their treatment between groups | 12 months
  The EORTC PATSAT-C33 questionnaire assesses the delivery of oncology care as a whole with a score from 1-5; the EORTC OUT-PATSAT7 is a complementary questionnaire to assess the delivery of ambulatory oncology care with a score from 1-5.
Patient satisfaction with their treatment between groups | 15 months
  The EORTC PATSAT-C33 questionnaire assesses the delivery of oncology care as a whole with a score from 1-5; the EORTC OUT-PATSAT7 is a complementary questionnaire to assess the delivery of ambulatory oncology care with a score from 1-5.
Patient satisfaction with their treatment between groups | 18 months
  The EORTC PATSAT-C33 questionnaire assesses the delivery of oncology care as a whole with a score from 1-5; the EORTC OUT-PATSAT7 is a complementary questionnaire to assess the delivery of ambulatory oncology care with a score from 1-5.
Quality of life adjusted years between groups | 18 months
  EuroQol-5 Dimension (EQ5D-3L) questionnaire, presented as 5-digit number
Cost of care between groups | End of study (18 months)
  The cost of the system will be estimated from the point of view of the health care institution by valuing the time of the medical and nursing staff and patient out-of-pocket expenses
Toxicity experienced during treatment between groups | 3 months
  National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)
Toxicity experienced during treatment between groups | 6 months
  National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)
Toxicity experienced during treatment between groups | 9 months
  National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)
Toxicity experienced during treatment between groups | 12 months
  National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)
Toxicity experienced during treatment between groups | 15 months
  National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)
Toxicity experienced during treatment between groups | 18 months
  National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE)
Relative Dose Intensity between groups | 3 months
  % doses received/dose planned
Relative Dose Intensity between groups | 6 months
  % doses received/dose planned
Relative Dose Intensity between groups | 9 months
  % doses received/dose planned
Relative Dose Intensity between groups | 12 months
  % doses received/dose planned
Relative Dose Intensity between groups | 15 months
  % doses received/dose planned
Relative Dose Intensity between groups | 18 months
  % doses received/dose planned
Budget Impact Analysis | After 2 years
  Cost of care for the population reached (actual population treated) on a national scale in Euros
Rate of prescription changes since initiation of oral therapy (whether change in usual treatment and oral therapy). | 3 months
Rate of prescription changes since initiation of oral therapy (whether change in usual treatment and oral therapy). | 6 months
Rate of prescription changes since initiation of oral therapy (whether change in usual treatment and oral therapy). | 9 months
Rate of prescription changes since initiation of oral therapy (whether change in usual treatment and oral therapy). | 12 months
Rate of prescription changes since initiation of oral therapy (whether change in usual treatment and oral therapy). | 15 months
Rate of prescription changes since initiation of oral therapy (whether change in usual treatment and oral therapy). | 18 months
Medication observance | 3 months
  Girerd questionnaire; score 0-6
Medication observance | 6
  Girerd questionnaire; score 0-6
Medication observance | 9 months
  Girerd questionnaire; score 0-6
Medication observance | 12 months
  Girerd questionnaire; score 0-6
Medication observance | 15 months
  Girerd questionnaire; score 0-6
Medication observance | 18 months
  Girerd questionnaire; score 0-6
Usability of the Thess monitoring patient interface for the collection of Patient Reported Outcomes | Month 18
  System Usability Scale questionnaire; score 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Fiteni, Principal Investigator — CHU de Nimes
Locations (6):
- France (6):
  - Centre Hospitalier Dubois Brive, Brive-la-Gaillarde
  - Chic Castres-Mazamet, Castres
  - Centre Hospitalier Emile ROUX, Le Puy-en-Velay
  - CHU de Nîmes, Nîmes
  - Institut cancerologie du Gard, Nîmes
  - Médipôle Lyon-Villeurbanne, Villeurbanne